CLINICAL TRIAL: NCT03078049
Title: Characteristics of Patients With Type 2 Diabetes Mellitus Receiving Treatment With Dapagliflozin Versus Sitagliptin: An Analysis of Commercial Claims and Linked Laboratory Data
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Optum, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00034
Record Dates: First submitted 2017-02-22; First posted 2017-03-13 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dapagliflozin: Patients taking dapagliflozin
- Sitagliptin: Patients take sitagliptin

SUMMARY:
Rationale: In order to compare the real-world use of commonly prescribed second-line oral diabetes therapies, real-world data comparing patients receiving treatment with dapagliflozin vs sitagliptin are needed, and limited resource use and cost data exist for patients initiating dapagliflozin in the real-world setting.

Objectives:

Primary: The primary objective of this study is to compare real-world health care resource utilization and costs following treatment with dapagliflozin versus sitagliptin. Secondary: The secondary objectives of this study are to assess clinical outcomes and treatment patterns among patients receiving treatment with dapagliflozin versus sitagliptin. Study Design: Retrospective cohort study. Target Subject Population: Patients receiving treatment with either dapagliflozin or sitagliptin will be evaluated.

Study Variable(s):

Primary Variables: Health care resource utilization and costs Secondary Variables: Demographics measured at the index date, Quan-Charlson Comorbidity score, measured during the baseline period, Agency for Healthcare Research and Quality (AHRQ)-based comorbidity measures, receipt of other antidiabetic medication classes during the baseline and follow-up periods, number and percentage of patients with a diagnosis of obesity during the baseline or follow-up periods, treatment patterns during the follow-up period (i.e., index dose, duration of treatment, discontinuation, adherence, receipt of additional antidiabetic medication classes), HbA1c outcomes (among subgroup of patients with linked laboratory data, sample size permitting), renal impairment, hypoglycemia as defined by a claims-based algorithm.

Statistical Methods: Initial analyses will be descriptive in nature and entail the tabular display of mean values, medians, ranges, and standard deviations of continuous variables of interest (e.g., patient age) and frequency distributions for categorical variables (e.g., sex, geographic location). Outcomes will be compared between patients receiving dapagliflozin versus sitagliptin using univariate tests. Propensity score matching will be undertaken to reduce bias in the comparison of patients receiving treatment with dapagliflozin versus sitagliptin. Following matching, demographics and baseline characteristics will be assessed using standardized differences to determine balance in the post-matched sample. Outcomes will be assessed using tests for paired data (paired t-tests, signed rank tests, McNemar's tests).

DETAILED DESCRIPTION:
Rationale: In order to compare the real-world use of commonly prescribed second-line oral diabetes therapies, real-world data comparing patients receiving treatment with dapagliflozin versus sitagliptin are needed, and limited resource use and cost data exist for patients initiating dapagliflozin in the real-world setting.

Objectives:

Primary:

The primary objective is to compare real-world health care resource utilization and costs following treatment with dapagliflozin versus sitagliptin.

Secondary:

The secondary objectives of this study are to assess the following real-world data among patients receiving treatment with dapagliflozin versus sitagliptin:

1. Patient demographic and baseline clinical and treatment characteristics
2. Treatment patterns, specifically dose at index date, duration of treatment, adherence, discontinuation, and receipt of additional antidiabetic agents
3. Clinical outcomes after treatment augmentation, including hypoglycemic events, renal impairment, and HbA1c

Study Design: Retrospective cohort study of commercial medical and pharmacy claims along with enrollment information and linked laboratory results between July 1, 2013 and April 30, 2016.

Target Subject Population: Patients receiving treatment with either dapagliflozin or sitagliptin will be evaluated in this analysis. The date of the first observed claim for either dapagliflozin or sitagliptin will define the index date. This study will use an intent- to-treat population, and patients will remain in their defined study cohort for the duration of the follow-up period, regardless of treatment changes. The baseline period will be defined as the 6 months' pre-index date, and the follow-up period will be defined as the 12 months' post-index date (inclusive of the index date). Patients will be required to have continuous health plan enrollment during the baseline and follow-up periods. Patients having at least one claim with a diagnosis of type 1 diabetes mellitus in the baseline period or gestational diabetes or evidence of pregnancy in the baseline or follow-up periods will be excluded from the study population. Furthermore, patients will be excluded from the analysis if they received a selective sodium glucose co-transporter-2 (SGLT-2) or dipeptidyl peptidase 4 (DPP-4) inhibitor during the baseline period. Patients receiving treatment with dapagliflozin will be matched on demographic, clinical, and economic characteristics to patients receiving treatment with sitagliptin using the 1:1 propensity score matching technique.

Study Variable(s):

Primary Variables: Health care resource utilization and costs

Secondary Variables:

1. Demographics measured at the index date
2. Quan-Charlson Comorbidity score, measured during the baseline period
3. Agency for Healthcare Research and Quality (AHRQ)-based comorbidity measures
4. Receipt of other antidiabetic medication classes during the baseline and follow-up periods.
5. Number and percentage of patients with a diagnosis of obesity during the baseline or follow-up periods
6. Treatment patterns during the follow-up period
7. HbA1c outcomes
8. Renal impairment
9. Hypoglycemia as defined by a claims-based algorithm

Statistical Methods:

All analyses including the assessment of patient demographics, patient characteristics, and health care utilization and costs will be descriptive in nature and entail the tabular display of mean values, medians, ranges, and standard deviations of continuous variables of interest and frequency distributions for categorical variables. Prior to matching, outcomes will be compared between patients receiving dapagliflozin versus sitagliptin using univariate tests. In Phase 2, propensity score matching will be undertaken to reduce bias in the comparison of patients receiving treatment with dapagliflozin versus sitagliptin. Following matching, demographics and baseline characteristics will be assessed using standardized differences to determine balance in the post-matched sample. Outcomes will be assessed using tests for paired data.

ELIGIBILITY:
Inclusion Criteria:

A prescription claim for either dapagliflozin or sitagliptin between on after January 1, 2014 (note: patients receiving dapagliflozin/metformin combination therapy (Xigduo), sitagliptin/metformin (Janumet/Janumet XR), or sitagliptin/simvastatin (Juvisync) will be included in the study population). The date of the first observed claim for either dapagliflozin or sitagliptin will define the index date.

Continuous medical and pharmacy benefits for a 6-month baseline period.

At least 1 diagnosis of T2DM in any position (ICD-9-CM and ICD-10-CM diagnosis codes are provided in accompanying Excel file) during the 6-month baseline period or during the 12- month follow-up period

Exclusion Criteria:

Receipt of either a SGLT-2 inhibitor or DPP-4 inhibitor during the 6-month baseline period.

A diagnosis of type 1 diabetes mellitus (T1DM) in any position during the baseline period.

A diagnosis of gestational diabetes mellitus (GDM) or pregnancy in any position during the 6-month baseline period or 12-month follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both Male and Female 18+
Sampling Method: Probability Sample
Enrollment: 11971 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Inpatient Stays | 6 months
  Number of patients with at least one hospital stay, number of unique stays and average length of stay.
Emergency Department Visits | 6 months
  Number of patients with at least one emergency department visit and number of emergency department visits.
Ambulatory visits (physician office visits and outpatient visits) | 6 months
  Number of patients with at least one visit and number of visits.
Other medical costs | 6 months
  Per-patient costs for medical services outside of inpatient hospitalization, emergency department visits, and ambulatory visits.
Total medical costs | 6 months
  Per-patient costs for all medical claims
Pharmacy Costs | 6 months
  Count of unique medications filled, count of medication fills, and per-patient costs for all pharmacy claims.
Total costs | 6 months
  Per-patient costs for all medical and pharmacy claims.

SECONDARY OUTCOMES:
Adherence | 6 months
  Proportion of days covered (PDC)
Discontinuation of index therapy | 6 months
  Discontinuation of index therapy will be defined as a gap in therapy of 60 days.
Persistence with index therapy | 6 months
  Persistence with therapy will be measured as days to therapy discontinuation (as defined above) or end of follow-up (in patients who do not discontinue) and the total number of prescription fills for the index therapy prior to discontinuation.
Follow-up within-class index medication switching | 6 months
  Patients with claims for other medications within the index class (use of other SGLT-2 agents for dapagliflozin patients and use of other DPP-4 agents for sitagliptin patients) during the follow-up period will be identified.
Follow-up index medication switching | 6 months
  Patients with claims for the other index medication (use of DPP-4 agents for dapagliflozin patients and use of SGLT-2 agents for sitagliptin patients) during the follow-up period will be identified.
Index dose | 6 months
  The dose of the index medication will be identified as 5mg or 10mg (dapagliflozin) or 25mg, 50mg, or 100mg (sitagliptin). Dose will be calculated by the drug strength x the quantity supplied/days supplied.
Index medication dose increase | 6 months
  Patients with a dose increase from the index dose for the index medication will be identified and the date of the first dose increase will be captured.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wittbrodt, PharmD, MPH, Study Director — AstraZeneca
Locations (1):
- Research Site, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
2 abstracts
  1 manuscript

REFERENCES:
- See also: ClinicalStudyReportSynopsis _D1690R00034 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14623&filename=ClinicalStudyReportSynopsis%20_D1690R00034.pdf